CLINICAL TRIAL: NCT02776020
Title: Non-invasive, Real-time Anesthetic Drug-monitoring System
Acronym: ADM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, ABECASSIS PHILIPPE, Head of women and obstetrics anesthesiology unit, Rambam Health Care Campus
Other Study IDs: 0347-15 RBM
Record Dates: First submitted 2016-05-09; First posted 2016-05-18 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Anesthesia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Propofol sedated patients: Women undergoing a short trans vaginal ovum retrieval (TVOR) will be sedated with propofol , and monitored non-invasively for changes in blood propofol concentration levels. Propofol dosages will be adapted according to patients vital signs and their reaction to noxious stimuli exerted during the trans vaginal ovum retrieval (TVOR) procedure, irrespective to the proposed study in which these participants undergo.Those changes of administered propofol dosages will be observed by the anesthetic drug monitor (ADM). Propfol is administered by the anesthesiologist in a routine manner and according to anesthesiologist discretion .
  Interventions: Device: CorrecDose Infrared Monitor

INTERVENTIONS:
Device: CorrecDose Infrared Monitor — The monitor is attached to patient's wrist and ear in order to measure changes in propofol concentrations in blood

SUMMARY:
The aim of this study is to determine efficacy of the "CorrecDose" device to continuously and non-invasively follow the changes in propofol concentrations in the participants' blood.

ELIGIBILITY:
Inclusion Criteria:

* Women who have signed Informed consent form
* Women undergoing Trans vaginal ovum retrieval (TVOR) for invitro fertilization (IVF) and will be sedated with propofol administered intravenos (IV)

Exclusion Criteria:

* Women with background diseases
* Women with chronic use of drug and medication
* Women with peripheral blood vessels problems
* Women with high blood pressure
* Women with body mass index (BMI) score over 35 or less than 18

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women undergoing propofol sedation while undergoing trans vaginal ovum retrieval (TVOR) for in vitro fertilization (IVF).
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-12 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Changes in Propofol Blood Levels | Half hour
  Graphic display on monitor of real-time changes

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Abecassis, MD, Principal Investigator — Rambam

IPD SHARING:
Plan to Share IPD: No